CLINICAL TRIAL: NCT02815969
Title: Exploring the Metabolic Profile of Neuroendocrine Tumors
Brief Title: The Indol Profile; Exploring the Metabolic Profile of Neuroendocrine Tumors
Status: Completed | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Other Study IDs: 201600496
Record Dates: First submitted 2016-06-21; First posted 2016-06-28 (Estimated); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Neuroendocrine Tumors
Keywords: neuroendocrine tumors; indol profile; catecholamines; LC-MS/MS
MeSH Terms: conditions — Neuroendocrine Tumors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Healthy volunteers: If no material of healthy volunteers of the SERT study can be used, then other matched volunteers are asked for a vena punction and urine collection
  Interventions: Other: vena punction
- Patients: Patients are asked for a vena punction and urine collection, if not already done because of medical care.
  Interventions: Other: vena punction

INTERVENTIONS:
Other: vena punction — vena punction and urine collection

SUMMARY:
This is an observational and exploratory study. Participants will be asked for a blood collection and a 24- hour collection of urine. The indol profile and levels of catecholamine and metabolites in PRP, as well as in 24- hour collection of urine will be measured with LC-MS/MS and analyzed.

DETAILED DESCRIPTION:
Rationale:

Neuro-endocrine neoplasms are a diverse group of tumors which encompasses heterogeneous clinical courses. Different NETs are characterized by differences in the synthesis, storage and release of biogenic amines and their metabolites, e.g. indoles, catecholamines and their metabolites. Clinical course, prognosis, and treatment are based, among others, on the origin of the primary tumor. Up to now it was only possible to measure metabolic output of NETs by serotonin in platelets and 5-HIAA in urine. Due to technical improvements we can now measure the complete metabolic pathway of serotonin in plasma and urine, which comprises tryptophan, 5-hydroxytryptophan, serotonin and 5-HIAA, the indol profile. Furthermore, levels of catecholamines and metabolites can now be analyzed in the same sample. This metabolic profiling could potentially lead to improved diagnosis and characterization of NET patients and possibly contribute to subsequent treatment consequences.

Therefore, we want to perform an exploratory study to measure the indol profile, catecholamines and metabolites in patients with NETs of different origin (foregut, midgut and hindgut) and assess differentiation of their metabolic profile.

Objective:

The aim of this study is to explore the added value of the indol profile in comparison to serotonin in platelets and 5-HIAA in urine for diagnosis and potentially management of neuroendocrine tumors including gastrinomas, pNETs and brochopulmonary NETs.

Design:

This is an observational and exploratory study. Participants will be asked for a blood collection and a 24- hour collection of urine. The indol profile and levels of catecholamine and metabolites in PRP, as well as in 24- hour collection of urine will be measured with LC-MS/MS and analyzed.

Study population:

In this study we will use PRP and a 24- hour collection of urine of 70 patients with a foregut NET, 70 patients with a midgut and/or hindgut NET and 70 matched healthy volunteers. Healthy volunteers are matched according to age and sex with the included patients. Matched controls already available in our data bank will be used from the earlier approved SERT study (NCT 01398306)

Main study parameters:

In this exploratory study we will measure the indol profile in patients with a foregut NET, mid- and hindgut NET, and healthy volunteers at the time of diagnosis and during follow up and treatment in plasma and urine.

In addition, levels of catecholamines and metabolites in these three groups will be determined.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

Patients with midgut NET already have blood collections and urinary collection as part of evaluation of their treatment. Only for patients with foregut NETs and some of the healthy volunteers one extra blood collection with a vena puncture will be taken. This gives a small risk of bruising. Furthermore a 24-hours collection of urine will be collected with a prescription to their diet 48 hours before the collection. This could give some distress.

ELIGIBILITY:
Inclusion criteria for all subjects:

* written informed consent
* age above 18 years

Inclusion criteria for patients with a NET: (one of these)

* histologically proven NET, with or without treatment for the NET
* a diagnosis made by a dedicated NET specialist based on a combination of physical symptoms and signs, imaging and laboratory values.

Inclusion criteria for healthy subjects:

- Matching in age (plus or minus 3 years) and sex with one of the included NET patients.

Data of healthy subjects could also be used from the SERT-study, if the subject meets the criteria mentioned above.

Exclusion criteria for all subjects:

* Use of drugs or food supplements that interact with the serotonin-metabolism; all serotonin re-uptake inhibitors, psychotrophic drugs, (other antidepressants; tricyclic antidepressants, MAO-inhibitors, mirtazapin, bupropion, venlafaxin, duloxetin, anxiolytic, antipsychotic and anticonvulsive drugs).
* Drug abuse in the last 8 weeks.
* Use of ≥ 14 alcoholic consumptions a week for women.
* Use of ≥ 21 alcoholic consumptions a week for men.

Exclusion criteria for healthy subjects:

* Having a neuroendocrine tumor or neuroendocrine carcinoma from any grade and location in present or in history.
* Having a malignancy.
* Having an auto-immune disease.
* Having an infection.
* Having renal impairment.
* Use of interferon.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with foregut NET, patients with a midgut and/or hindgut NET, and healthy volunteers. All patients will be included in one of the groups by a dedicated NET doctor based on a combination of physical symptoms and signs, laboratory values, imaging and histology.
Sampling Method: Probability Sample
Enrollment: 210 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2019-08 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
indol profile; 5-HTP, Serotonin, 5-Hydroxyindolacetic acid, Tryptophan in platelet rich plasma | at one visit
  indol profile in platelet rich plasma

SECONDARY OUTCOMES:
catecholamines; L-DOPA, Dopamine, Norepinephrine, Epinephrine, -Methoxytyramine, Normetanephrine, Metanephrine in platelet rich plasma | at one visit
  catecholamines in platelet rich plasma
indoles and catecholamines; L-DOPA, 5-HTP, Dopamine, Norepinephrine, Epinephrine, 3-Methoxytyramine, Normetanephrine, Metanephrine, Serotonin, 5-Hydroxyindolacetic acid | at one visit
  indoles and catecholamines in urine

CONTACTS AND LOCATIONS:
Overall Officials: A. M.E. Walenkamp, MD, PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No